CLINICAL TRIAL: NCT00090038
Title: A Multicenter Study to Evaluate the Effect of Rituximab (IDEC-102) on Primary Humoral Response, Recall Response, and Maintenance of Acquired Immunity to Specific Antigens
Brief Title: Effect of Rituximab on Immunological Recall Response to Specific Antigens in the Treatment of Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-12
Record Dates: First submitted 2004-08-23; First posted 2004-08-24 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rituximab
  Interventions: Drug: rituximab
- 2 (No Intervention): No drug

INTERVENTIONS:
Drug: rituximab — Dose, schedule,and duration specified in protocol
  Arms: 1

SUMMARY:
The purpose of this study is to provide treatment for patients who have relapsed Non-Hodgkin's lymphoma (NHL) or refractory NHL, and to test the immunity of study subjects after receiving four treatments with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Signed IRB-approved informed consent.
* Age >/=40 years.
* Men and women of reproductive potential who are following accepted birth control methods.
* Histologic confirmation of low-grade or follicular, B-cell NHL prior to study entry.
* Relapsed (maximum of 5 relapses) or refractory, low-grade or follicular, CD20+,B-cell NHL.
* WHO performance status </= 2.
* Expected survival >/= 1 year.
* Acceptable hematologic status, liver function, renal function, and pulmonary function.
* Patients must be recovered from all nonhematological toxicities associated with prior surgery, radiation treatments, chemotherapy, biological therapy, bone marrow transplant, investigational drugs, or immunotherapy.
* Known history of tetanus toxoid immunization or positive tetanus titer at the screening visit.

Exclusion Criteria:

* Active autoimmune disease.
* Exposure to rituximab within 12 months prior to Day 1.
* Chemotherapy within 3 months prior to Day 1.
* Previous immunization with tetanus toxoid within 2 years prior to Day 1.
* Previous exposure to KLH.
* Receipt of intravenous or intramuscular immunoglobulin (IVIG or IMIG) within 30 days of Day 1.
* Known history of hepatitis or other hepatic disease, HIV infection, or AIDS.
* Current use (including "recreational use") of any illicit drugs or history of drug or alcohol abuse within the 5 years prior to Day 1.
* Prior diagnosis of aggressive NHL or mantle-cell lymphoma.
* Chronic lymphocytic leukemia (CLL).
* Small lymphocytic lymphoma (IWF A) with peripheral blood lymphocyte count > 5,000 cells/mm3.
* History of other primary malignancy, with the exception of squamous cell carcinoma or basal cell carcinoma of the skin, in situ carcinoma of the cervix, or treated prostate cancer for which the subject has not been disease free for at least 3 years.
* Serious nonmalignant disease (e.g., congestive heart failure, hydronephrosis); active, uncontrolled bacterial, viral, or fungal infection; or any other condition that would compromise protocol objectives in the opinion of the investigator and/or sponsor.
* Known allergies or contraindications to tetanus toxoid or KLH.
* Known allergy to shellfish.
* Presence of protein-losing enteropathy.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1.
* Participation in another clinical study with an investigational agent or device within the last year. The subject cannot participate in any other clinical study with an investigational agent or device during the course of this study.
* Pregnant or lactating female subjects

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2003-10; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine whether treatment with rituximab causes a clinically significant effect on immunological recall response to tetanus vaccine in NHL patients | 8.5 months after treatment

SECONDARY OUTCOMES:
To determine whether NHL patients can mount a primary response to KLH after treatment with rituximab | 8.5 months after treatment
To determine whether NHL subjects treated with rituximab experience clinically significant changes in antibody titers to a panel of specific antigens | 8.5 months after treatment

CONTACTS AND LOCATIONS:
Locations (45):
- United States (7):
  - USC KECK School of Medicine, Los Angeles, California
  - Radiant Research, Honolulu, Hawaii
  - Carle Clinic Association, Urbana, Illinois
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - University of Pittsburth Cancer Centers, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Research Site, Graz, Austria
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (4):
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Strasbourg
- Germany (9):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Frankfurt
  - Research Site, Giessen
  - Research Site, Hamburg
  - Research Site, Koblenz
  - Research Site, Mainz
  - Research Site, Mutlangen
  - Research Site, Tübingen
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
- Russia (5):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Research Site, Stockholm, Sweden
- Turkey (Türkiye) (3):
  - Research Site, Gaziantep
  - Research Site, Izmir
  - Research Site, Kayseri
- United Kingdom (4):
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Manchester
  - Research Site, Sheffield